CLINICAL TRIAL: NCT00026403
Title: A Phase II Study of Gemcitabine, Cisplatin and Radiation Therapy in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9942; NCI-2012-02426 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000069026 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- radiotherapy + gemcitabine + cisplatin (Experimental): Patients undergo radiotherapy once daily five days a week for 5.5 weeks. Patients receive gemcitabine IV over 30 minutes followed by cisplatin IV over 1 hour twice a week for the first 3 weeks of radiotherapy. Beginning 4 weeks after the completion of radiotherapy, patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for a total of 3 courses in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline, at completion of radiotherapy, at completion of chemotherapy, and 3 months after completion of therapy.
  Patients are followed every 3 months for 2 years and then every 6 months for 1 year.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of gemcitabine, cisplatin, and radiotherapy, in terms of 1-year survival, in patients with locally advanced pancreatic cancer.
* Determine the toxicity of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo radiotherapy once daily five days a week for 5.5 weeks. Patients receive gemcitabine IV over 30 minutes followed by cisplatin IV over 1 hour twice a week for the first 3 weeks of radiotherapy. Beginning 4 weeks after the completion of radiotherapy, patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for a total of 3 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at completion of radiotherapy, at completion of chemotherapy, and 3 months after completion of therapy.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 20-47 patients will be accrued for this study within 12-28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable adenocarcinoma of the pancreas
* No cystadenocarcinoma of the pancreas or pancreatic tumors of neuroendocrine origin
* Prior subtotal resection or gross residual disease

  * No microscopic residual disease only
* No metastatic disease outside of planned study radiotherapy field

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to maintain adequate oral nutrition
* No significant infection
* No other medical condition that would preclude study
* No other malignancy within the past 5 years except non-melanoma skin cancer
* No significant nausea or vomiting

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior or concurrent biologic therapy

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy that would overlap planned study radiotherapy fields

Surgery:

* See Disease Characteristics
* At least 21 days since prior laparotomy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-09; Primary Completion 2007-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
overall survival | 12 months

SECONDARY OUTCOMES:
quality of life | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Haddock, MD, Study Chair — Mayo Clinic
Locations (26):
- United States (25):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Haddock MG, Swaminathan R, Foster NR, Hauge MD, Martenson JA, Camoriano JK, Stella PJ, Tenglin RC, Schaefer PL, Moore DF Jr, Alberts SR. Gemcitabine, cisplatin, and radiotherapy for patients with locally advanced pancreatic adenocarcinoma: results of the North Central Cancer Treatment Group Phase II Study N9942. J Clin Oncol. 2007 Jun 20;25(18):2567-72. doi: 10.1200/JCO.2006.10.2111. PMID 17577035
- [Result] Haddock MG, Swaminathan R, Alberts SR, et al.: Gemcitabine (Gem), cisplatin (Cis) and radiation therapy (RT) for patients with locally advanced pancreatic adenocarcinoma (ACA): a North Central Cancer Treatment Group (NCCTG) phase II study. [Abstract] J Clin Oncol 22 (Suppl 14): A-4121, 343s, 2004.